CLINICAL TRIAL: NCT03528356
Title: The Impact of Dietary Counseling on the Efficacy of Tooth Bleaching: a Randomized Controlled Trial
Brief Title: Impact of Dietary Counseling on Efficacy of Tooth Bleaching
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPGO026
Record Dates: First submitted 2018-05-07; First posted 2018-05-17 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Tooth Discoloration
MeSH Terms: conditions — Tooth Discoloration | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular diet (Placebo Comparator)
  Interventions: Behavioral: Regular diet
- White diet (Experimental)
  Interventions: Behavioral: Regular diet

INTERVENTIONS:
Behavioral: Regular diet — Patients will not receive any information regarding their usual diet. They will simply perform home dental bleaching.

SUMMARY:
The aim of this study will be to evaluate if subjects submitted to a white diet counseling during home dental bleaching will present better results than subjects that maintained their usual diets. Forty patients will be divided into two groups and randomly allocated to each group: usual diet (control) or white diet, avoiding dye-containing food and beverages. patients will be assessed through a food frequency questionnaire and color measurement using a spectrophotometer at baseline and six months after bleaching.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 18 or higher;
* Central incisors with shade A2 or darker

Exclusion Criteria:

* Undergone previous dental bleaching procedures;
* Under orthodontic treatment;
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-30 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Tooth color | 6 months
  Will be assessed using a spectrophotometer

SECONDARY OUTCOMES:
Food frequency questionnaire | 6 months
  Patients will respond to a 30 item questionnaire regarding their daily diet. A Food Frequency Questionnaire (FFQ) was constructed to evaluate the consumption of chromogenic food and beverage of patients in the last year. A list of 54 foods and beverages that, according to the literature, have the potential to cause some kind of extrinsic pigmentation, was elaborated. In each food of beverage, the individual will be asked if he consumed in the last year and if the answer is yes, the consumption frequency (0 to 10 times) per unit of time (day, week, month or year). In addition, each individual will answer regarding the amount relative to the mean portion, half of the mean portion, or twice of the mean portion. The size of the mean portions will be considered by calculating the mean of each food consumed. The home measure for the mean portion will be based on the Table of Evaluation of Food Consumption in Home Measures (Pinheiro et al. 2000).

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Univeristy of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No